CLINICAL TRIAL: NCT00805116
Title: Whale Oil Versus Cod Liver Oil in Rheumatoid Arthritis
Brief Title: Marine Oils and Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment to slow, most patients to well for treatment
Sponsor: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Responsible Party: Principal Investigator, Marian Kjellevold, Head of Research, National Institute of Nutrition and Seafood Research, Norway
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1523 Hvalolje (NIFES); REK VEST 257.07; NSD 17989
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Cod Liver Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Whale blubber oil
  Interventions: Dietary Supplement: Whale blubber oil
- 2 (Active Comparator): Cod liver oil
  Interventions: Dietary Supplement: Cod liver oil

INTERVENTIONS:
Dietary Supplement: Whale blubber oil — 15 ml/day for 4 months, divided on dosage morning and evening, orally.
  Arms: 1
Dietary Supplement: Cod liver oil — 15 ml/day for 4 months, divided on dosage morning and evening, taken orally
  Arms: 2

SUMMARY:
NSAIDS are associated with adverse GI effects and COX-2 inhibitors have cardiovascular risk. Long-term oral supplementation with fish oil reduce e.g. joint pain in rheumatoid arthritis (R.A) patients, with reduced need for NSAIDS, in addition to being cardioprotective. The aim is to investigate if 4 month supplementation of 15 ml/day of whale blubber oil compared with cod liver oil reduce the intensity of joint pain in patients with R.A (primary outcome). Patients are assessed at inclusion and after study (4 months) during routine polyclinical visit. Patients are called for interview after 6 and 12 weeks. Secondary outcomes are e.g. morning stiffness, quality of life and functional level

DETAILED DESCRIPTION:
Not relevant

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients according to American College of Rheumatology criteria (with active disease and in remission). Intensity of joint pain last week (30 mm or more on 100 mm Visual analogue scale). Stable use of DMARDS and no corticosteroid injections last 4 weeks before study and during study.

Exclusion Criteria:

* Non-Norwegian speaking/reading or not understanding study design or non-compliance. Pregnant/lactating women. Bleeder disease, known HIV or hepatitis, medication with Marevan (blood thinner). Not willing or possible to stop taking regular omega-3 supplements during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To detect a difference in 10 mm on visual analogue scale (intensity of joint pain last week) between the two treatment groups | At study end (4 months)

SECONDARY OUTCOMES:
To detect a group difference in morning stiffness last week in minutes (720 min = 12 hours are limit for duration of morning stiffness recorded) | Study end (4 months)
To detect a difference between groups in quality of life using SF-36 | Study end (4 months)
To see a group difference in functional level using MHAQ | Study end (4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Livar Frøyland, Dr, Study Director — NIFES